CLINICAL TRIAL: NCT00731770
Title: TITLE: Double-blinded, Double-dummy, Study Comparing Fluticasone-salmeterol to Placebo in Patients With COPD and Associated Poor Sleep or Daytime Somnolence.
Brief Title: Comparing Fluticasone-salmeterol in Chronic Obstructive Pulmonary Disease (COPD) and Sleep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Timothy Craig, Timothy Craig, D.O., Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 29024
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: COPD
Keywords: COPD; sleep; daytime somnolence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disorders of Excessive Somnolence | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo, then Advair 250- matched (Placebo Comparator): 1 puff bid Placebo for two weeks followed by a 4 week washout period with placebo. After the washout period, they then received Advair 250- matched 1 puff bid for two weeks.
  Interventions: Drug: Advair 250; Drug: Placebo- matched
- Advair 250, then Placebo- matched (Active Comparator): 1 puff bid Advair 250 for two weeks followed by a 4 week washout period with placebo. After the washout period, they then received Placebo- matched 1 puff bid for two weeks.
  Interventions: Drug: Placebo; Drug: Advair 250 - matched

INTERVENTIONS:
Drug: Advair 250 — 1 puff bid inhaled
  Other Names: fluticasone/salmeterol 250/50
  Arms: Placebo, then Advair 250- matched
Drug: Placebo- matched — 1 puff bid inhaled
  Arms: Placebo, then Advair 250- matched
Drug: Placebo — Placebo 1 puff bid inhaled
  Arms: Advair 250, then Placebo- matched
Drug: Advair 250 - matched — i puff bid inhaled
  Other Names: fluticasone/salmeterol 250/50
  Arms: Advair 250, then Placebo- matched

SUMMARY:
Fluticasone (Advair), an inhaled corticosteroid and salmeterol, a long-acting beta agonist, are approved for use in the management of COPD. Fluticasone/salmeterol has been shown to significantly improve forced expiratory volume (FEV1) and decrease COPD symptoms (Calverley et al. 2003, 2007). Inhaled corticosteroids have been shown to decrease frequency of COPD exacerbations (Gartlehner et al. 2006) and long acting bronchodilators demonstrated a reduction in dyspnea, increased airflow and reduction in hyperinflation in patients with symptomatic COPD (Ramirez-Venegas et al. 1997). Specifically, salmeterol has also been shown to have a positive effect on symptoms and health status of patients with COPD when added to usual treatment (Stockley et al. 2006).

Previous research of subjects from our group with asthma has shown salmeterol to be associated with sustained improvements in morning peak expiratory flow (PEF), protection from nighttime lung function deterioration and improvement in patient perception of sleep (Wiegand et al. 1999). This study has not been performed in patients with COPD nor has the effect of salmeterol with fluticasone on sleep quality been assessed.

AIM: The aim of this study is to determine the effect of fluticasone/salmeterol on sleep quality in patients with COPD and to compare efficacy of Advair 250 compared to placebo on sleep.

The hypothesis is that there would be a significant improvement in sleep quality when patients are placed on fluticasone/salmeterol as compared to placebo.

DETAILED DESCRIPTION:
RATIONALE:

Chronic obstructive pulmonary disease (COPD) is a term that describes a disease state in which there is chronic irreversible airflow limitation. It has been well documented that patients with COPD have disturbed sleep. Certain published reports suggest that more than 50% of COPD patients have sleep complaints (George et al., Drugs, 2003). These patients are found to have sleep onset latency and poor sleep maintenance. While their sleep disturbance may be explained in part by side effects of medications, it could also be a result of nocturnal gas exchange abnormalities (Knutty 2004). In COPD there is worsening hypoxemia and hypercapnia during sleep, particularly rapid eye movement (REM) sleep, and sleep disturbance seems to be worse with more severe COPD. It is commonly believed that optimizing medical management of the disease is important in improving the sleep quality of these patients and thus leading to improved quality of life.

Fluticasone, an inhaled corticosteroid and salmeterol, a long-acting beta agonist, are approved for use in the management of COPD. Fluticasone/salmeterol has been shown to significantly improve FEV1 and decrease COPD symptoms (Calverley et al. 2003, 2007). Inhaled corticosteroids have been shown to decrease frequency of COPD exacerbations (Gartlehner et al. 2006) and long acting bronchodilators demonstrated a reduction in dyspnea, increased airflow and reduction in hyperinflation in patients with symptomatic COPD (Ramirez-Venegas et al. 1997). Specifically, salmeterol has also been shown to have a positive effect on symptoms and health status of patients with COPD when added to usual treatment (Stockley et al. 2006).

Previous research of subjects from our group with asthma has shown salmeterol to be associated with sustained improvements in morning PEF, protection from nighttime lung function deterioration and improvement in patient perception of sleep (Wiegand et al. 1999). This study has not been performed in patients with COPD nor has the effect of salmeterol with fluticasone on sleep quality been assessed.

AIM:

The aim of this study is to determine the effect of fluticasone/salmeterol on sleep quality in patients with COPD and to compare efficacy of Advair 250 compared to placebo on sleep.

The hypothesis is that there would be a significant improvement in sleep quality when patients are placed on fluticasone/salmeterol as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate to severe COPD as per GOLD criteria
2. Insomnia, poor sleep, non-restorative sleep or daytime sleepiness by history
3. Age 45 to 75 years, male or female
4. FEV1 below 80% of predicted using CRAPO
5. FEV1/FVC < 70% predicted
6. Past or present tobacco smoker
7. Female patients must be postmenopausal for 1 year or be willing to use birth control or abstain from sex.

Exclusion Criteria:

1. Asthma
2. Use of oral or injectable corticosteroids within 2 months
3. Previous diagnosis of sleep disorder breathing (sleep apnea, narcolepsy, etc.)
4. Lung or heart disease except for COPD
5. Deviated nasal septum, nasal polyps or anatomic obstruction of the nose
6. Obesity defined as BMI >30kg/m2
7. Inability to tolerate or history of allergy to long acting beta agonist or inhaled corticosteroid therapy.
8. Inability to complete a 2 week run-in with albuterol prn as only therapy
9. Use of narcotics, sleep aids, sedating antihistamines, sedatives, MAO Inhibitors, and other medications known to affect daytime somnolence or sleep quality
10. Excessive use of alcohol or use of "recreational drugs"
11. Use of narcotics, sleep aids, sedatives or sedating antihistamines.
12. Night shift workers
13. Women who are breast feeding or pregnant.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Craig, DO, Principal Investigator — Penn State University
Locations (1):
- Penn State Universuty, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Advair 250, Then Palcebo- Matched: 1 puff bid Advair 250 for two weeks followed by a 4 week washout period with placebo. After the washout period, they then received Placebo- matched 1 puff bid for two weeks.
Period: Overall Study
Arm/Group | Placebo, Then Advair 250- Matched | Advair 250, Then Palcebo- Matched
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the Institution and no baseline data are available for reporting. Sincere efforts were made to obtain the data, but were unsuccessful.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Advair 250- Matched | Advair 250, Then Placebo- Matched | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical — data was not analyzed and is no longer available for analysis
Sex: Female, Male — data was not analyzed and is no longer available for analysis
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Aim of This Study is to Determine the Effect of Fluticasone/Salmeterol on Sleep Quality in Patients With COPD and to Compare Efficacy of Advair 250 Compared to Placebo on Sleep.
Time Frame: 1 year
Population: Th PI has left the Institution and no outcome data are available for reporting. Sincere efforts were made to obtain the data, but were unsuccessful.
Arm/Group | Placebo, Then Advair 250- Matched | Advair 250, Then Palcebo- Matched
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Daytime Somnolence
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Placebo, Then Advair 250- Matched | Advair 250, Then Placebo- Matched
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Placebo: 1 puff bid Placebo for two weeks followed by a 4 week washout period with placebo. After the washout period, they then received Advair 250- matched 1 puff bid for two weeks.
- Advair 250: 1 puff bid Advair 250 for two weeks followed by a 4 week washout period with placebo. After the washout period, they then received Placebo- matched 1 puff bid for two wee
Arm/Group | Placebo | Advair 250
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Th PI has left the Institution and no outcome data are available for reporting. Sincere efforts were made to obtain the data, but were unsuccessful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No